CLINICAL TRIAL: NCT01203540
Title: Evaluation of the Effect and Tolerance of Preservative Free NAAGA on the Inflammatory Component and Symptoms of Dry Eye Syndrome in Allergic Conjunctivitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Collaborators: Samil Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NBKE_SNUBH&BM_01; LT0455-IST-01/10
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naaga in ABAK system (Experimental)
  Interventions: Drug: NAABAK eyedrops
- Saline solution (Placebo Comparator)
  Interventions: Drug: Saline eyedrops

INTERVENTIONS:
Drug: NAABAK eyedrops
  Arms: Naaga in ABAK system
Drug: Saline eyedrops
  Arms: Saline solution

SUMMARY:
Multicentre, Double blind, Randomized, Comparative Study(comparing N-acetyl-aspartyl-glutamic acid(NAAGA) in Abak preservative free device versus SALINE in Abak preservative free device.

Evaluation of the effects and safety of NAABAK® through inflammation markers and symptoms in patients with allergic conjunctivitis and dry eye syndrome after 3 months treatment.

The patients will attend 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* Patients with dry eye syndrome in allergic conjunctivitis

Exclusion Criteria:

* Severe dry eye syndrome
* Severe ocular pathology

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2010-10; Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Boramae Medical Center, Seoul